CLINICAL TRIAL: NCT05954091
Title: A Phase 1, Open-label Study of OH2, an Oncolytic Virus, Administered by Intratumoral Injection in Patients with Advanced/Metastatic Solid Tumors
Brief Title: OH2 Administered by Intratumoral Injection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-007
Record Dates: First submitted 2023-06-05; First posted 2023-07-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- OH2 Injection (Experimental): Subjects will get OH2 injection every two weeks, and up to 8mL for each treatment. There will have three virus titers: 1×10^6 CCID50/mL, 5×10^6 CCID50/mL, 1×10^7 CCID50/mL.
  Interventions: Drug: OH2 Injection

INTERVENTIONS:
Drug: OH2 Injection — OH2 injection will be given intratumorally, and Q2W.
  Other Names: BS001

SUMMARY:
This study will be a Phase 1, multi-center, open-label, dose escalation followed by the recommended phase 2 dose (RP2D) expansion study to characterize safety, tolerability, biodistribution, virus shedding and preliminary efficacy of intratumoral injection of OH2 in patients with locally advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
Eligible patients are those who have measurable solid tumors as detected by CT or MRI that have persisted, recurred, or metastasized despite therapy. Part 1 and Part 2 Cohort A will include patients who have solid tumors with cutaneous/subcutaneous tumor lesions, such as melanoma, cutaneous squamous cell carcinoma, and cutaneous/subcutaneous metastasis from pancreatic cancer, colorectal cancer, breast cancer, etc. Part 2 Cohort B will include patients who have visceral tumors. Patients who were previously treated with IMLYGIC (Talimogene laherparepvec, T-Vec) but did not achieve an optimal response to T-Vec are eligible to receive OH2 if otherwise per protocol (refer to Section 5 for detailed enrollment criteria). The study will be conducted in 2 parts as described below. Both parts will consist of a screening period of up to 28 days, a treatment period and a follow-up period (safety and long-term follow up). Treatment period of Part 1 will include an initial treatment period (namely DLT (dose-limiting toxicity) observation period, 3 doses of OH2) and an optional extended treatment period (repeated every 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years old
2. Subject must have histologically- or cytologically-confirmed diagnosis of unresectable locally advanced or metastatic melanoma, pancreatic cancer, liver metastases from colorectal cancer, breast cancer, and other solid tumors. (Part 1 and Part 2 Cohort A will include patients who have solid tumors with cutaneous/subcutaneous tumor lesions, such as melanoma, cutaneous squamous cell carcinoma, and cutaneous/subcutaneous metastasis from pancreatic cancer, colorectal cancer, breast cancer etc. Part 2 Cohort B will include patients who have visceral tumors.)
3. Subject has measurable disease as determined by RECIST version 1.1. At least 1 lesion must be suitable for intratumoral (IT) injection. Lesions for injection must be ≥ 10 mm and ≤ 60 mm in longest diameter.
4. Subjects who have progressed on or are ineligible for available standard therapy are eligible for this trial after the last dose of the previous treatment which is ≥ 4 weeks or 5 half-lives (if required) before the first dose of study treatment. Note: patients who have previously been treated with IMLYGIC (Talimogene laherparepvec, T-Vec) are eligible after discontinuing the last dose of previous T-Vec treatment for ≥ 12 weeks before first dose of study treatment.
5. Subject has a predicted life expectancy ≥ 12 weeks.
6. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. A female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

   * Not a woman of childbearing potential (WOCBP) OR
   * WOCBP who agrees to use an acceptable form of birth control method, including:

   abstinence, hormonal contraception for at least 3 months in combination with a barrier method, intrauterine device (placement at least 3 months prior to screening), cervical cap, condoms with contraceptive gel/foam/cream, or surgical sterilization (tubal ligation at least 6 months prior to screening or partner who had a vasectomy at least 6 months prior to screening).
8. Female subject must agree not to breastfeed starting at screening, throughout the study period and 180 days after the final study IP administration.
9. Female subject must not donate ova starting at screening, throughout the study period and for 180 days after the final study IP administration.
10. Male subject must agree to remain abstinent or use a condom throughout the study period and for 180 days after the final study IP administration.
11. Male subject with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 180 days after the final study IP administration.
12. Male subject must not donate sperm during the treatment period and for at least 180 days after the final study IP administration.
13. Subject must be willing and able to comply with the study requirements including prohibited concomitant medication restrictions.
14. Subject agrees not to participate in another interventional study while receiving study IP.
15. Subject has the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subject has ongoing toxicity ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 2 attributable to prior antineoplastic therapies considered clinically significant determined by the Investigator.
2. Subject has had major surgery ≤ 4 weeks of screening.
3. Subject is concurrently participating in another interventional study or has received an investigational product < 4 weeks or 5 half-lives (if required) prior to first IP administration.
4. Subject with symptomatic central nervous system (CNS) metastases, except patients with CNS lesions that have been treated and have no evidence of progression in the brain on CT/MRI for ≥ 3 months and have been off steroids for at least 4 weeks prior to first IP administration.
5. Subject with active autoimmune disease requiring systemic therapy within past 2 years. (e.g., systemic lupus erythematosus, Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, hypophysitis, etc.). The following are exceptions to this criterion:

   * Subject with vitiligo or alopecia
   * Subject with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Childhood asthma that has resolved
   * Any chronic skin condition that does not require systemic therapy
   * Type 1 diabetes mellitus ※Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
6. Subject with another malignancy that currently requires treatment.
7. Subject with tumors encasing major vascular structures such as the carotid artery, tumors adjacent to vital neurovascular structures or tumors in locations that are at high risk for AEs or otherwise not considered appropriate for IT injection.
8. Subject with inadequate organ and marrow functions meeting any of the below criteria:

   * with ongoing continuous supportive treatment
   * Leukocytes < 3000/μL
   * Absolute neutrophil count < 1500/μL
   * Platelets < 100,000/μL
   * Hemoglobin (Hgb) < 9 g/dL
   * International normalized ratio (INR) > 1.5 × ULN and/or activated partial thromboplastin time (aPTT) > 1.5 × institutional normal limits, except for patients in Group B (Visceral Lesions) escalation and expansion groups where INR and aPTT must be normal
   * Total Bilirubin (TBL) > 1.5 × institutional normal limits (subjects with known Gilbert syndrome who are excluded if TBL > 3.0 × institutional normal limits or direct bilirubin > 1.5 × institutional normal limits)
   * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) > 3.0 × institutional normal limits. Subjects with tumors in the liver AST and ALT > 5 × institutional normal limits.
   * Albumin < 3.0 g/dL
   * Creatinine > 1.5 × institutional normal limits
9. Subject with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of first administration of study IP. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
10. Subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, any form of substance abuse or psychiatric illness/social situations that would limit compliance with study visits or requirements, or a condition that could invalidate communication with the Investigator.
11. Subject is known to be positive for human immunodeficiency virus, hepatitis B surface antigen, hepatitis B core immunoglobulin or immunoglobulin G (IgG) antibody, or hepatitis C (IgG or ribonucleic acid (RNA) test) indicating acute or chronic infection. HbsAg positive subject should further undergo hepatitis B virus (HBV) DNA titer detection. For HCV antibody positive subject, further HCV RNA testing is required. However, subject with the following conditions can be included in this study: Hepatitis B surface antigen (HBsAg) is negative; if HBcAb is positive, HBV-DNA (HBV deoxyribonucleic acid) < 200 IU/mL (or 1000 copies/mL).
12. Subject has a history of moderate to severe ascites, clinically significant and/or rapidly accumulating ascites, bleeding esophageal varices, hepatic encephalopathy, or pericardial and/or pleural effusions related to liver insufficiency within 6 months of screening. Mild ascites that does not preclude safe IT injection of OH2 is allowed.
13. Subject has a clinically significant abnormal electrocardiogram (ECG) at screening.
14. Subject has symptomatic cardiovascular disease within the preceding 12 months unless cardiology consultation and clearance has been obtained for study participation, including but not limited to the following: significant coronary artery disease (e.g., requiring angioplasty or stenting), acute myocardial infarction or unstable angina pectoris < 3 months prior to screening, uncontrolled hypertension, clinically significant arrhythmia, or congestive heart failure (New York Heart Association grade ≥ 2).
15. Subject who has a history of bleeding diathesis, are on anti-coagulation therapy, or have abnormal coagulation-fibrinolytic parameters (e.g., activated partial thromboplastin time (APTT), prothrombin time (PT), thrombin time (TT), and platelet count).
16. Subject has medical conditions that predispose the subject to untoward medical risk in the event of volume loading (e.g., intravenous fluid bolus infusion), tachycardia, or hypotension during or following treatment with OH2.
17. Subject has a known or suspected hypersensitivity to OH2 or any components of the formulation used, including prior adverse reaction to vaccinia (e.g., as smallpox vaccine).
18. Subject has had previous exposure with OH2.
19. Active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis).
20. Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Event (AE) and Serious Adverse Event (SAE) | Through study completion, an average of about 1 year(a maximum treatment duration of one year)
  Toxic reactions according to the NCI-CTCAE 5.0 grading standard that occur within 3 weeks from the first administration, are judged to be drug-related by the investigator, and meet the non-hematological toxicity and hematological toxicity conditions specified in the clinical protocol
Maximum tolerated dose (MTD) | up to 1 year
  To estimate the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of OH2

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 1 year
  Determination of the ORR is calculated based on the proportion of patients achieving complete response (CR) or partial response (PR) using the RECIST v1.1 and modified WHO response criteria as assessed.
Disease control rate (DCR) | up to 1 year
  DCR is defined as the percentage of participants with a best overall response of CR, PR, or stable disease (SD).
Biological activity | up to 1 year
  Granulocyte macrophage colony stimulating factor (GM-CSF) mRNA expression in fine needle aspirate (FNA)(Only for Part 1)
Biodistribution | 3 months
  OH2 DNA copy in blood and urine
Viral shedding | 3 months
  OH2 DNA copy in swab of surface of injected lesion

IPD SHARING:
Plan to Share IPD: No